CLINICAL TRIAL: NCT05246488
Title: Reliability and Validity Study of the American Orthopedic Foot and Ankle Society Midfoot Scale
Brief Title: Validation of the American Orthopedic Foot and Ankle Society Midfoot Scale
Status: Completed | Type: Observational
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Yasemin Şahbaz, doctoral lecturer, University of Beykent
Other Study IDs: UBeykent-2
Record Dates: First submitted 2022-02-08; First posted 2022-02-18 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Foot
Keywords: foot; validity; reliability
MeSH Terms: interventions — Visual Analog Scale

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: American Orthopedic Foot and Ankle Association Midfoot Scale, Foot and Ankle Ability Measure/FAAM, SF-12 Quality of Life Scale, Visual Analog Scale (VAS) — All participants will receive two assessments, 7 days apart. After the demographic data of the patients are recorded with the form prepared by us, they will be evaluated with the AOFAS Midfoot Scale, Foot and Ankle Ability Measure/FAAM, SF-12 Quality of Life Scale, Visual Analogue Scale (VAS).

SUMMARY:
Today, one of the frequently used scales in the evaluation of foot problems is the American Orthopedic Foot and Ankle Association Scale. AOFAS has been prepared with the American society in mind and its original version is in English. This limits the application of AOFAS to non-English speaking patients. The aim of study is to investigate the cross-cultural adaptation, reliability and validity of the Turkish version of the AOFAS Midfoot Scale.

DETAILED DESCRIPTION:
Foot and ankle disorders are the most common disorders affecting the musculoskeletal system and greatly affect patients' quality of life. Due to the complex anatomy and function of the foot, accurate diagnosis is an important clinical problem, making it difficult to locate the source of pain with routine clinical examination. There are many scales developed in academic studies or clinical practices to help diagnose or to evaluate foot-ankle diseases and accompanying symptoms and conditions.

The American Orthopedic Foot and Ankle Score is one of the widely used clinical outcome measures specifically designed to examine the foot and ankle. It consists of four grading systems, with each system set up to study a different anatomical area. These are the ankle-hindfoot, midfoot, hallux-metatarsophalangeal-interphalangeal, and smaller metatarsophalangeal-interphalangeal joints. The scale, which includes objective and subjective items, was developed to assess pain, function and smoothness. The original version of AOFAS is in English, which limits its application to non-English speaking patients. Some parts of AOFAS have been translated and culturally adapted into Turkish, Italian, German and Persian. The Turkish translation and cultural adaptation of AOFAS was completed only for the Ankle-Back Foot Scale out of the four rating systems. In this study, aimed to investigate the translation, cross-cultural adaptation, reliability and validity of the Turkish version of the AOFAS Midfoot Scale.

Translation and Cultural Adaptation Translation and cross-cultural adaptation of the AOFAS Midfoot Scale. It will be carried out in 5 stages, in line with the stages proposed by . In the first stage, the scale will be translated into Turkish independently by 2 Turks who have a good command of English. In the second stage, both translations will be compared in terms of conceptual errors and consistency by a bilingual translator. In the third stage, after the agreement is reached on the first Turkish translation, 2 native English speakers with a good command of Turkish will separately translate the completed Turkish translation into English. The purpose of this work will not be disclosed to both translators and they will not have access to the original English version. In the fourth stage, the translated version of the AOFAS Midfoot Scale will be compared with the original English version of the AOFAS Midfoot Scale by a committee of a methodologist, a linguist and 4 translators. The committee will be asked to evaluate the 4 translations and compare the inconsistencies and finalize them for approval.

Evaluations All participants will receive two assessments, 7 days apart. After the demographic data of the patients are recorded with the form prepared by us, they will be evaluated with the AOFAS Midfoot Scale, Foot and Ankle Ability Measure/FAAM, SF-12 Quality of Life Scale, Visual Analogue Scale.

AOFAS Midfoot The validity and reliability scale prepared by the American Orthopedic Foot-Ankle Association consists of three sub-dimensions. Evaluations in pain, function, smoothness sections and total scores range from 0 to 100 points. High scores indicate severe deformity and low scores indicate milder deformity.

Foot and Ankle Usability Measure FAAM is a 29-item questionnaire including 21-item activities of daily living and 8-item sports subscales. The maximum score of the 5-point Likert-type scale is 84 for activities of daily living and 32 points for the sports subscale. The total score varies between 0-100. A higher score corresponds to a higher level of function for both subscales. The validity and reliability study of the scale was conducted.

S-12 Quality of Life Scale The SF-12 Quality of Life Scale is a scale to evaluate quality of life by taking 12 questions from 8 different sub-dimensions of the SF-36 Quality of Life Scale. The shorter the scale, the easier it is in terms of applicability. The scale has a different scoring method than the SF-36. In the short form SF-12, physical and mental component summary scores are calculated as sub-dimensions. The total score of the physical and mental component summary of the scale varies between 0-100. An increase in the score indicates well-being, and a decrease indicates a state of disability. The validity and reliability study of the scale was conducted.

Visual Analog Scale, participants are asked to select the point where they feel pain on a 10-centimeter horizontal line. 0 - no pain, 10 - unbearable pain. Pain conditions are evaluated separately at night, during activity and at rest.

Statistical Method SPSS 25.0/Statistical Package for Social Sciences Inc; Chicago, IL, USA statistical program will be used in all statistical analyses. For all variables, mean±standard deviation and percent values will be presented within the scope of descriptive statistics. In the evaluation of test results, the level of significance will be considered as p<0.05. Measurement properties for the examined scales will be analyzed in terms of internal consistency, test-retest reliability, construct validity, floor and ceiling effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Patients who were operated for Lisfranc and midfoot tarsometatarsal pathologies
* Patients who are followed up and treated in the orthopedic service
* Having the ability to read and write Turkish
* Those who agreed to participate in the study

Exclusion Criteria:

* patients under the age of 18
* Patients with nerve injury and peripheral neuropathy, sensory loss, neuromuscular pathological findings, infection, acute fractures in the lower extremities, and acute rheumatic disease
* Patients who are followed up and treated in external centers

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 40 patients who applied to Bakirkoy Dr. Sadi Konuk Training & Research Hospital Orthopedics and Traumatology Clinic between 15.02.2022 and 15.08.2022 and were operated due to midfoot pathologies will be included in the study.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
American Orthopedic Foot and Ankle Association Midfoot Scale | through study completion, an average of 6 months
  The validity and reliability scale prepared by the American Orthopedic Foot-Ankle Association consists of three sub-dimensions. Evaluations in pain, function, smoothness sections and total scores range from 0 to 100 points. High scores indicate severe deformity and low scores indicate milder deformity.
Foot and Ankle Usability Measure | through study completion, an average of 6 months
  FAAM is a 29-item questionnaire including 21-item activities of daily living and 8-item sports subscales. The maximum score of the 5-point Likert-type scale is 84 for activities of daily living and 32 points for the sports subscale. The total score varies between 0-100. A higher score corresponds to a higher level of function for both subscales. The validity and reliability study of the scale was carried out.

SECONDARY OUTCOMES:
S-12 Quality of Life Scale | through study completion, an average of 6 months
  Developed by Ware et al., the SF-12 Quality of Life Scale is a scale to evaluate quality of life by taking 12 questions from 8 different sub-dimensions of the SF-36 Quality of Life Scale. The shorter the scale, the easier it is in terms of applicability. The scale has a different scoring method than the SF-36. In the short form SF-12, physical (SF12-PCS) and mental (SF12-MCS) component summary scores are calculated as sub-dimensions. The total score of the physical and mental component summary of the scale varies between 0-100. An increase in the score indicates well-being, and a decrease indicates a state of disability. The validity and reliability study of the scale was carried out.
Visual Analog Scale (VAS) | through study completion, an average of 6 months
  Participants are asked to select the point where they feel their pain on a 10-centimeter (cm) horizontal line. 0 - no pain, 10 - unbearable pain. Pain conditions are evaluated separately at night, during activity and at rest.

CONTACTS AND LOCATIONS:
Overall Officials: assis.prof. Altuğ Duramaz, Principal Investigator — ISTANBUL BAKIRKOY DR. SADİ KONUK EDUCATION AND RESEARCH HOSPITAL; as.dr. Alican Koluman, Principal Investigator — ISTANBUL BAKIRKOY DR. SADİ KONUK EDUCATION AND RESEARCH HOSPITAL; as.dr. Mehmet Utku Çiftçi, Principal Investigator — ISTANBUL BAKIRKOY DR. SADİ KONUK EDUCATION AND RESEARCH HOSPITAL; assis.prof. Tansu Birinci, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Beykent University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kitaoka HB, Alexander IJ, Adelaar RS, Nunley JA, Myerson MS, Sanders M. Clinical rating systems for the ankle-hindfoot, midfoot, hallux, and lesser toes. Foot Ankle Int. 1994 Jul;15(7):349-53. doi: 10.1177/107110079401500701. PMID 7951968
- [Background] Celik D, Malkoc M, Martin R. Evidence for reliability, validity and responsiveness of Turkish Foot and Ankle Ability Measure (FAAM). Rheumatol Int. 2016 Oct;36(10):1469-76. doi: 10.1007/s00296-016-3485-4. Epub 2016 May 2. PMID 27136921
- [Background] Celik D, Coban O. Short Form Health Survey version-2.0 Turkish (SF-36v2) is an efficient outcome parameter in musculoskeletal research. Acta Orthop Traumatol Turc. 2016 Oct;50(5):558-561. doi: 10.1016/j.aott.2016.08.013. Epub 2016 Nov 17. PMID 27866914
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Garcia Jimenez R, Garcia-Gomez FJ, Noriega Alvarez E, Calvo Moron C, Martin-Marcuartu JJ. Hybrid imaging in foot and ankle disorders. Rev Esp Med Nucl Imagen Mol (Engl Ed). 2018 May-Jun;37(3):191-202. doi: 10.1016/j.remn.2017.10.003. Epub 2017 Dec 6. English, Spanish. PMID 29221678
- [Background] Reed MD, Van Nostran W. Assessing pain intensity with the visual analog scale: a plea for uniformity. J Clin Pharmacol. 2014 Mar;54(3):241-4. doi: 10.1002/jcph.250. Epub 2014 Jan 23. No abstract available. PMID 24374753
- [Background] Analay Akbaba Y, Celik D, Ogut RT. Translation, Cross-Cultural Adaptation, Reliability, and Validity of Turkish Version of the American Orthopaedic Foot and Ankle Society Ankle-Hindfoot Scale. J Foot Ankle Surg. 2016 Nov-Dec;55(6):1139-1142. doi: 10.1053/j.jfas.2016.06.001. Epub 2016 Sep 7. PMID 27614824
- [Background] Leigheb M, Janicka P, Andorno S, Marcuzzi A, Magnani C, Grassi F. Italian translation, cultural adaptation and validation of the "American Orthopaedic Foot and Ankle Society's (AOFAS) ankle-hindfoot scale". Acta Biomed. 2016 May 6;87(1):38-45. PMID 27163894
- [Background] Vosoughi AR, Roustaei N, Mahdaviazad H. American Orthopaedic Foot and Ankle Society ankle-hindfoot scale: A cross-cultural adaptation and validation study from Iran. Foot Ankle Surg. 2018 Jun;24(3):219-223. doi: 10.1016/j.fas.2017.02.007. Epub 2017 Feb 17. PMID 29409212
- [Background] Kostuj T, Krummenauer F, Schaper K, Stief F, Zettersten K, Baums MH, Meurer A, Lieske S. Analysis of agreement between the German translation of the American Foot and Ankle Society's Ankle and Hindfoot Scale (AOFAS-AHS) and the Foot Function Index in its validated German translation by Naal et al. (FFI-D). Arch Orthop Trauma Surg. 2014 Sep;134(9):1205-10. doi: 10.1007/s00402-014-2046-0. Epub 2014 Jul 11. PMID 25012530